CLINICAL TRIAL: NCT01938105
Title: Preoperative Concurrent Chemoradiotherapy Combined With Nimotuzumab Injection for Locally Advanced Cervical Cancer: a Phase II Study
Brief Title: Preoperative Chemoradiotherapy Combined With Nimotuzumab for Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Principal Investigator, Heming Lu, Associate Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WJPMF-2013-428-2081
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Cervical cancer; Nimotuzumab; Intensity-modulated radiation therapy; Concurrent chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab+chemoradiotherapy (Experimental)
  Interventions: Other: Nimotuzumab+chemoradiotherapy

INTERVENTIONS:
Other: Nimotuzumab+chemoradiotherapy — Nimotuzumab 200mg per week will be administered concurrent with platinum-based chemotherapy and intensity-modulated radiation therapy. After the preoperative treatment, patients will be assessed for tumor response and operability. For those who are considered to be candidates for operation, radical surgery will be performed.
  --------------------------------------------------------------------------------

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of preoperative nimotuzumab injection combined with concurrent chemoradiotherapy for initially inoperable, locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell cervical cancer
* Stages IB2-IIIB according to FIGO Staging System
* Age:18-75
* ECOG<2
* Normal bone marrow function
* Initial assessed and considered not candidates for operation
* Signed study-specific consent form

Exclusion Criteria:

* Pregnant or lactating women
* Patients with other malignancies
* Patients who received radiotherapy or chemotherapy previously
* Presence of uncontrolled life-threatening illness
* Allergy to platinum or monoclonal antibody

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Treatment related toxicities | at 1 year
  Acute and chronic toxicities.
Tumor response after preoperative treatment | assessed at 4-5 weeks after the completion of preoperative treatment

SECONDARY OUTCOMES:
Progression-free survival | at 1 year
Overall survival | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heming Lu, MS, Study Chair — People's Hospital of Guangxi Zhuang Autonomous Region; Heming Lu, MS, Principal Investigator — People's Hospital of Guangxi Zhuang Autonomous Region; Yun Mo, MS, Principal Investigator — People's Hospital of Guangxi Zhuang Autonomous Region
Locations (1):
- People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi, China